CLINICAL TRIAL: NCT04191005
Title: Efficacy of Platelet-Rich Plasma Therapy for Androgenetic Alopecia: A Systematic Review and Meta-analysis
Acronym: PRP IN AGA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jasim Mohammed Alshammari (Other)
Responsible Party: Sponsor-Investigator, Jasim Mohammed Alshammari, director, Assiut University
Organization: Assiut University (Other)
Other Study IDs: PRP in Androgentic Alopecia
Record Dates: First submitted 2019-12-04; First posted 2019-12-09 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
assess the literature on PRP outcomes for AGA, with a focus on specific clinical outcomes in a comparative view, in accordance with PRISMA statement for reporting this meta-analysis

DETAILED DESCRIPTION:
Androgenic alopecia (AGA) also known as androgenetic alopecia or male pattern baldness, is a common disorder that affects both men and women. Is one of the commonest reasons for dermatological consultation worldwide (1). It is characterized by progressive hair loss, especially of scalp hair, and has distinct patterns of loss in women versus men. AGA is an age-dependent disorder characterized by patterned hair loss. Based on the few prevalence data available, Know that by the age of 30 years about 30% of men will have AGA and that this will rise to about 50% by the age of 50 years and as many as 90% in their lifetime (2) , Although prevalence increases with age in all populations, thinning can begin as early as puberty (3). The hair thinning begins between the ages of 12 and 40 years in both sexes and approximately half the population expresses this trait to some degree before the age of 50 years (4). Androgentic alopecia is familial with a complex polygenic mode of inheritance (5) . Polymorphism of the androgen receptor gene, the 5 a reductase gene and 2 other, as yet unidentified genes on chromosomes 3 and 21 have been all been associated with premature balding (6). There is a family tendency towards androgenetic alopecia and it is thought to have a polygenic mode of inheritance. Alopecia causes major discomfort due to altered appearance with significant implications in daily living and possible leading to depression and anxiety symptoms with a significantly higher prevalence in AGA female compared with male subjects (7). Pathophysiology upon entry of testosterone into the hair follicle via dermal papilla's capillaries, binding occurs to the androgen receptors (ARs) either directly or after its conversion to dihydrotestosterone (DHT) (8). AGA is known to be mediated by the conversion of circulating androgens into DHT within the hair follicle .In the hair follicle cells, testosterone converts into the biologically more active metabolite; DHT, which is considered the key androgen required for the induction of AGA (9). This conversion is catalyzed by the enzyme 5α-reductase type-II. Binding of androgens to their ARs leads to conformational change of the AR-androgen complex which is then transported into the nucleus where it can bind to DNA which has distinctive binding sites: In most men, AGA involves the fronto temporal area and the vertex, following a pattern corresponding to the Hamilton- Norwood scale (10). In women, typically three patterns have been 1-Diffuse thinning of the crown region with preservation of the frontal hairline 2-Thinning and widening of the central part of the scalp with breach of frontal hairline, 3- Thinning associated with bitemporal recession (Hamilton-Norwood type, diagnostic evaluation form for AGA, including history, clinical evaluation like scalp and hair examination and diagnostic techniques and test (Pull test, Wash test), and clinical documentation . AGA can be treated medically, surgically or cosmetically (11) The most recommended treatment for AGA is composed of local minoxidil, hormonal therapy such as local and oral antiandrogens (12).

Platelet-rich plasma (PRP) is used as an innovative therapy in diverse fields including dentistry, surgery, orthopedics, dermatology and aesthetics (13). Currently, PRP preparation systems have FDA clearance for use in bone grafts and operative Orthopedics but off-label purposes such as for hair restoration have become increasingly common. PRP is a rich source of growth factors such as insulin-like growth factor 1 (IGF-1), platelet-derived growth factor (PDGF), transforming growth factor-b (TGF-b), vascular endothelial growth factor (VEGF), epidermal growth factor (EGF) and fibroblast growth factor (FGF) which together can stimulate cell survival, proliferation, differentiation, vascularization and angiogenesis (14). Application of these growth factors to dermal papilla (DP) cells can lead to the initiation and prolongation of anagen phase in the hair follicle. Alpha granules within the platelets contain the growth factors and facilitate release at high concentrations, when the PRP preparation is activated. PRP is produced through cell separation by commercial kits or manual methods using a laboratory centrifuge and then injected into androgen-dependent areas of the scalp ( 15). With more hair restoration clinics choosing to offer PRP therapy, data on treatment efficacy have begun to accumulate. The AGA application remains in the early stages as treatment protocols are still being refined. At this time, PRP has been used in combination with hair transplant surgery and as an injectable therapy alone. Furthermore, diverse methods are reported as activators can be used to stimulate growth factor release; additional components such as leukocytes and dalteparin and protamine micro particles may be included to boost results; and quantity and frequency of treatments have varied widely (16).

The conduction of a meta-analysis provides systematic assessment of previous research studies to derive conclusions about that body of research. Outcomes from a meta-analysis may include a more precise estimate of the effect of treatment than any individual study .

ELIGIBILITY:
Inclusion Criteria:

* 1- Search for and assess studies comparing local injections of PRP compared to any control for AGA.

  2- Studies to be included in this review will be matched with predetermined criteria according to the PICOS (patients, intervention, comparator, outcomes, and study design) approach.

  3- These studies must include patients with any age and stage of AGA , with a minimum of 10 patients, a minimum of 3 months follow -up.

  4- Local injection of any autologous of PRP preparation into the scalp of AGA patients for treatment of AGA.

  5- Measure the efficacy of PRP therapy for treatment of AGA.

Exclusion Criteria:

1. Review, expert opinion, comments, letter to editor, case reports, studies on animals, conference reports will be excluded from the study.
2. Studies of other types of alopecia (i.e., alopecia areata or cicatricial alopecia) or studies with less than 10 patients, follow up less than 3 months or with no outcome reported, will be excluded from the study.

   -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data will be abstracted from every study in the form of a risk estimate and its 95% confidence interval (C1). Pooled risk estimate will be obtained by weighting each study by the inverse variance of the effect measure on algorithmic scale. This approach to pooling the results assumes that the study population being compared are similar and hence correspond to affixed effect analysis. The validity of pooling the risk estimate will be tested (test of homogeneity) using the chi-square test. A violation of this test implies that the studies being grouped differ from one another. In the presence of significant heterogeneity of the effect measure among studies being compared,
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-01-07 (Estimated); Primary Completion 2020-01-20 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
number of hair per square centimeter | one year
  measure the number of hairs per square centimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Manal mohamed Darwish, ass.professor, Study Director — community medicine; Rofaida refaat Shahata, doctor, Principal Investigator — dermatology
Locations (1):
- Assiut University, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Severi G, Sinclair R, Hopper JL, English DR, McCredie MR, Boyle P, Giles GG. Androgenetic alopecia in men aged 40-69 years: prevalence and risk factors. Br J Dermatol. 2003 Dec;149(6):1207-13. doi: 10.1111/j.1365-2133.2003.05565.x. PMID 14674898
- [Background] Varothai S, Bergfeld WF. Androgenetic alopecia: an evidence-based treatment update. Am J Clin Dermatol. 2014 Jul;15(3):217-30. doi: 10.1007/s40257-014-0077-5. PMID 24848508
- [Background] Norwood OT. Male pattern baldness: classification and incidence. South Med J. 1975 Nov;68(11):1359-65. doi: 10.1097/00007611-197511000-00009. PMID 1188424
- [Background] Stevens J, Khetarpal S. Platelet-rich plasma for androgenetic alopecia: A review of the literature and proposed treatment protocol. Int J Womens Dermatol. 2018 Sep 21;5(1):46-51. doi: 10.1016/j.ijwd.2018.08.004. eCollection 2019 Feb. PMID 30809579
- See also: Stevens, J., & Khetarpal, S. (2018). Platelet-rich plasma for androgenetic alopecia: A review of the literature and proposed treatment protocol. International journal of women's dermatology. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Platelet-rich+plasma+for+androgenetic+alopecia%3A+A+review+of+the+literature+and+proposed+treatment+protocol+Stevens+J%2C